CLINICAL TRIAL: NCT06144736
Title: PRIMETEST II - Phase II Trial to Prospectively Test New Predictors for Recurrence in Patients With Clinical Stage II A/B Seminoma Treated With RA-RPLND
Brief Title: PRIMETEST II - Clinical Stage II A/B Seminoma Treated With RA-RPLND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2256
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Seminoma
Keywords: seminoma; low volume metastases; clinical stage IIA/B
MeSH Terms: conditions — Seminoma | interventions — Etoposide; Bleomycin

STUDY DESIGN:
Intervention Model Description: The patients are classified as "low risk" or "high risk" for recurrence upon study enrollment. "Low risk" patients undergo a robot-assisted retroperitoneal lymph node dissection and metastasis resection (RA-RPLND) in a unilateral dissection field ("template") without adjuvant therapy. "High risk" patients also undergo a retroperitoneal lymph node dissection and metastasis resection in a unilateral dissection field, but additionally have the option to receive adjuvant therapy with one cycle of PEB two to four weeks after the RA-RPLND.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low risk (Experimental): Criteria for "low risk":
  * Absence of "high risk" criteria
  * Previous carboplatin therapy post orchiectomy
  * Exclusion of malignancy in the RPLND histology
  Interventions: Procedure: Robot-assisted retroperitoneal lymph node dissection
- High risk (Experimental): Criteria for "high risk":
  * Clinical stage II at initial diagnosis
  * Primary tumor > 4 cm
  * Infiltration of the "rete testis" in the primary tumor
  Interventions: Procedure: Robot-assisted retroperitoneal lymph node dissection; Drug: Adjuvant therapy with one cycle of cisplatin, etoposide and bleomycin

INTERVENTIONS:
Procedure: Robot-assisted retroperitoneal lymph node dissection — Robot-assisted, if possibe ipsilateral nerve-sparing, retroperitoneal lymph node dissection and metastasis resection in a unilateral dissection field ("template")
Drug: Adjuvant therapy with one cycle of cisplatin, etoposide and bleomycin — The patient is given the option for an adjuvant therapy with one cycle of cisplatin, etoposide and bleomycin two to four weeks after RA-RPLND
  Arms: High risk

SUMMARY:
PRIMETEST II is an interventional study involving low-volume metastatic seminoma. It explores a novel approach using robot-assisted primary retroperitoneal lymph node dissection, aiming to reduce long-term side effects and improve quality of life. By identifying factors predicting cancer recurrence, the study hopes to tailor treatments for better outcomes. The approach could potentially spare patients from chemotherapy induced long-term side effects while maintaining excellent survival rates, presenting a promising shift in testicular cancer care for this specific patient group.

DETAILED DESCRIPTION:
Testicular cancer stands as the most prevalent cancer among young men, boasting a highly favorable prognosis characterized by almost unaltered long-term survival even in advanced stages. However, traditional treatments like chemotherapy and radiation are linked to significant long-term toxicity and increased rates of secondary malignancies. Particularly, late toxicities, mainly cardiovascular, substantially diminish overall survival by approximately 6-7 years. To circumvent unnecessary acute and long-term toxicities associated with radiation or chemotherapy, it's crucial to explore alternative therapeutic avenues through personalized, less toxic approaches.

Building upon the hypothesis-generating PRIMETEST I study, PRIMETEST II is a single-arm, non-randomized prospective study. It aims to explore novel and personalized predictive parameters for recurrence following a robot-assisted primary retroperitoneal lymph node dissection (pRA-RPLND) in patients with clinical stage IIA/B seminoma (involving low-volume metastatic disease up to 5 cm). These patients represent a rare subgroup among testicular cancer patients, making a randomized comparison of treatment options impractical due to their low prevalence. The overarching goal is to reduce long-term toxicity in this young cohort of cancer patients and enhance their quality of life through personalized clinical and molecular predictions.

PRIMETEST I has indicated that pRA-RPLND in patients with clinical stage IIA/B seminoma led to a 70% recurrence-free survival at 32 months' follow-up. These findings suggest that pRA-RPLND could serve as an alternative to standard therapies (chemotherapy, radiotherapy) for a highly selective group of patients, effectively preventing excessive toxicity. PRIMETEST I has already identified several potential factors that predict which patients are more likely to benefit from surgical therapy alone.

In the novel prospective setting of PRIMETEST II, the study tests the identified predictive factors for recurrence. Patients exhibiting presumably low-risk features (about 70% of patients) will continue with surgery alone. Those with a presumed higher risk of recurrence will undergo robot-assisted surgery and have the option of receiving adjuvant treatment (one cycle of cisplatin, etoposide, and bleomycin). The primary endpoint is a three-year recurrence-free survival, estimated to exceed 90%. Additional objectives include exploring new predictors of recurrence at both molecular and clinical levels by analyzing serum and tissue samples from the primary tumor and metastases.

This innovative approach anticipates that 70% of patients will avoid long-term toxicity and experience excellent recurrence-free survival rates comparable to standard chemotherapy or radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pure seminomatous testicular germ cell tumor
* Presence of iliac or retroperitoneal lymph node metastasis detected in contrast-enhanced CT or MRI, classified as local or unilaterally regional
* Maximum extent of lymph node metastasis (LN-M) singular or multiple, with a maximum size of 5 cm in transverse CT diameter (UICC IIB)
* Patients with an elevation in HCG after orchiectomy at the time of staging examination can be included if the directly preoperatively determined HCG does not exceed 5 IU/L.

Patients can be included in the following scenarios:

* Initial diagnosis of a tumor in UICC stage IIA/IIB
* Recurrence of a tumor in clinical stage (CS) I under active surveillance
* Recurrence of a CS I tumor after adjuvant therapy with carboplatin mono

Exclusion Criteria:

* LN-M with a transverse diameter >5 cm in CT (UICC IIC)
* Other metastases than LN-M (UICC III)
* The patient received a different chemotherapy than described above
* The patient underwent retroperitoneal radiotherapy
* The patient is in a reduced general condition or has a life-threatening illness
* The patient has a psychiatric illness
* Evidence of non-seminomatous germ cell tumor components in the RPLND histology
* Complete resection cannot be ensured due to previous surgeries
* In the "high risk" group: Contraindications to cisplatin, etoposide, or bleomycin (severe liver insufficiency, severe kidney insufficiency, severe lung insufficiency, hypersensitivity, severe bone marrow depression, profound hearing impairments)

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | at least 5 years
Time to progression | from intervention to progression assessed up to 5 years
Complications | intra- and perioperative
  Intraoperative Adverse Incident Classification (EAUiaiC) by the European Association of Urology ad hoc Complications Guidelines Panel, Clavien-Dindo
Quality of life | baseline and yearly, up to 5 years
  EORTC QLQ-C30 and QLQ-TC26
Mental health | baseline and yearly, up to 5 years
  Questionnaire
Rate of retrograde ejaculation | postoperative assessment yearly, up to 5 years
Validation of microRNA-371 | Day before surgery, day 3-5 after surgery and in case of adjuvant therapy 3 days from last drug application
  Measurements of the biomarker microRNA-371
Analysis of molecular characteristics | after study recruitment completion
  Measurements still not specified

CONTACTS AND LOCATIONS:
Overall Officials: Yue Che, Principal Investigator — University Hospital of Düsseldorf
Locations (1):
- University Hospital of Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided